CLINICAL TRIAL: NCT04190719
Title: Patient Empowerment for Major Surgery Preparation @ Home: Multimodal Prehabilitation in Major Elective Surgery
Brief Title: Patient Empowerment for Major Surgery Preparation @ Home
Acronym: Paprika
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: EIT Health (Other); Hospital Clinic of Barcelona (Other); Universitätsklinikum Köln (Other); University Clinical Centre, Gdansk (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 38RC19.182
Record Dates: First submitted 2019-12-03; First posted 2019-12-09 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2020-11

CONDITIONS: Urologic Diseases; Cardiovascular Diseases; Thoracic Diseases; Orthopedic Disorder; Gastrointestinal Disease
MeSH Terms: conditions — Urologic Diseases; Cardiovascular Diseases; Thoracic Diseases; Musculoskeletal Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: Interventional group: Patients with Paprika program Historical group: Patients with same characteristics operated in 2018-2019
Masking Description: Paprika program will be proposed to all eligible patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paprika group (Experimental): Patients coming for elective major surgery will participate to Paprika program
  Interventions: Other: multimodal prehabilitation
- Historical group (No Intervention): Patients previously operated with same characteristics

INTERVENTIONS:
Other: multimodal prehabilitation — Paprika prehabilitation program content: patients will have choices for each activity. Messages and motivation will be reinforced by using a mobile app or leaflet advices, according to patient's preferences.
  * Physical activity promotion by discovering ebike, personalised gymnastics and encouragement to increase the number of daily steps of patients, measured by a wristband and a mobile App
  * An individualized nutritional optimization plan with dietary advices and protein supplementation (if necessary).
  * Psychological support will be proposed through auto-hypnosis sensibilisation or management of stress with Cognitive Behavior Stress Management technics
  Arms: Paprika group

SUMMARY:
Non-randomized monocentric open cohort study vs historical comparative group testing the efficacy of a multimodal prehabilitation program (based on physical activity, nutritional support and mental preparation) for unfit patients based on nutrition, physical activity and mental preparation in reducing postoperative complications in elective major surgery

DETAILED DESCRIPTION:
Prehabilitation programs essentially based on physical activity improvement may reduce postoperative complications after major surgery. We hypothesize that a multimodal program based on physical activity, nutritional support and mental preparation may not only improve postoperative recovery and reduce costs but also improve health status beyond postoperative period.

Non-randomized monocentric open cohort study vs historical comparative group testing the efficacy of a multimodal prehabilitation program for unfit patients based on nutrition, physical activity and mental preparation in reducing postoperative complications in elective major surgery.

Other outcomes will be measured : length of hospital stay, hospital readmissions, direct costs, health status at 1 and 6 months.

Moreover, the feasibility and adherence of Paprika program will be evaluated. Inter-data centres relating to the implementation of the same prehabilitation program will be compared with the consortium Paprika (Hospital Clinic of Barcelona, University of Cologne, University of Gdansk)

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible to elective major surgery (digestive, orthopedic, vascular-thoracic, urologic)
* Age > 70 years and/or American Society of Anesthesiologists (ASA) score 3-4
* or Unfit patient according to appropriate scores (Two among 3 scores (HAD, Physical activity score, nutritional score) below threshold). Unfit patients will be defined by at least 2 criteria if 'YES' answers: Physical activity: Less than 50% of WHO recommendations = less than 5000 steps/day or less than 75 min moderate activity/week or less than 12 min moderate activity/day Yes/No Malnutrition: BMI < 20 kg/m2 if < 70 years (or <22 if >70y) = undernutrition Yes/No or BMI>25 kg/m2 (= overweight to obesity) or Loss of appetite? Mental evaluation HAD (Hospital Anxiety and Depression) >8 for A or D score Yes/No
* Diagnosis:

Elective major surgery (digestive, orthopedic, vascular-thoracic, urologic)

- Regulatory aspects: Be legally able to give consent Patient affiliated to social security

Exclusion Criteria:

* Planned surgery (less than 4 weeks at inclusion)
* Urgent surgery
* Patient with, at baseline, good to excellent physical, nutritional, mental status as defined by appropriate scores.
* Patient considered not eligible to this program for physical or psychological reasons by the surgeon or the anesthetist
* Persons referred in Articles L1121-5 to L1121-8 of the French code of public health (this corresponds to all persons protected: pregnant or parturient women, breastfeeding mothers, persons deprived of liberty by judicial or administrative decision, persons subject to a legal protection measure).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative complications at Day-30 | at Day-30 post surgery
  Rate of postoperative complications at Day-30 classified following the standards of the European Society of Anaesthesiology and European Society of intensive Care Medicine.

SECONDARY OUTCOMES:
Number and severity of postoperative complications | within 30 days post surgery
  Number and severity of postoperative complications using Dindo-Clavien classification within 30 days
Length of stay (ICU and Hospital) | within 30 days post surgery
  Length of ICU stay and Length of hospital stay
Hospital readmission | within 30 days post surgery
  Hospital readmission within 30 days
Direct cost | interventional group: 1 month-cost before surgery+1 month-post surgery / Control group: 1 month-cost post-surgery
  Valuation in euros of the direct cost from a 1-month hospital point of view (duration and type of stay, acts, GHM...) by integrating for the intervention group the cost of the pre-habilitation program. Care consumption at 6 months from a social security perspective (Probabilistic Matching National Health Data System)--> comparison of direct costs for the Prehab sessions (professional caregivers and materials costs) versus complication costs of control group
Physical activity health status | a baseline, presurgery and 6 months post surgery
  Health status based on physical activity score:GPAQ and DASI scores
Nutritional health status | at baseline, 1 month and 6 months
  Nutritional health status based on weight, appetite and ingesta measurements
Psychological health status | at baseline, 1 month and 6 months
  Psychological health status based on HAD, Perceived Stress Scale scores
Number of patient participation to program in relation to the number of eligible patients | During Paprika inclusion period
  Number of patient participation to program in relation to the number of eligible patients to assess faisability
Ratio patient participation to each session | During Paprika 1 month-sessions
  Ratio patient participation to each session to assess faisability and limitation to participation
Comparison with other centers | through study completion, an average of 1 year
  Comparison will be done with other cohorts using Paprika program (Barcelona, Gdansk and Köln) on common outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Albaladejo, Prof., Principal Investigator — CHU Grenoble Alpes
Locations (1):
- Centre Hospitalier Universitaire Grenoble Alpes, La Tronche, France

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared with Barcelona, Köln and Gdansk: all collected IPD
Supporting Information: CSR
Time Frame: Data will be available at the end of the study: starting July 2021
Access Criteria: IPD will be shared with other sites in order to compare results coming from common questionnaires and data. Statistical analyses will be performed for Grenoble site separately and pooled with the other sites in a second step.

REFERENCES:
- [Result] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682
- [Result] Barberan-Garcia A, Ubre M, Pascual-Argente N, Risco R, Faner J, Balust J, Lacy AM, Puig-Junoy J, Roca J, Martinez-Palli G. Post-discharge impact and cost-consequence analysis of prehabilitation in high-risk patients undergoing major abdominal surgery: secondary results from a randomised controlled trial. Br J Anaesth. 2019 Oct;123(4):450-456. doi: 10.1016/j.bja.2019.05.032. Epub 2019 Jun 25. PMID 31248644